CLINICAL TRIAL: NCT00243308
Title: A Phase 2, Multicentre, Double-Blind, Placebo-Controlled, Dose Escalating Trial of the Safety, Pharmacokinetics, and Biological Activity of 3 Consecutive Daily Doses of Serp-1 When Added to Conventional Therapy in Patients With Acute Coronary Syndromes (Non ST-Elevation Myocardial Infarction and/or Unstable Angina)
Brief Title: Serp-1 for the Treatment of Acute Coronary Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Third dose group not recruited due to slow enrollment.
Sponsor: Viron Therapeutics Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Serp-1-01-002
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Unstable Angina; Coronary Atherosclerosis; Coronary Restenosis
Keywords: Anti-inflammatory agents; unstable plaque; acute coronary syndrome
MeSH Terms: conditions — Angina, Unstable; Coronary Artery Disease; Coronary Restenosis; Acute Coronary Syndrome

INTERVENTIONS:
Drug: Serine proteinase-1 (Serp-1)

SUMMARY:
Males and females aged 18-80 years who present with ACS (unstable angina and non ST-elevation MI) defined as one or more episodes of angina lasting at least 5 minutes in the last 24 hours before admission and greater than 0.05 mV of presumed new ST-segment depression in at least 2 contiguous ECG leads OR, angina and per confirmatory angiogram, has been scheduled for percutaneous coronary angioplasty. The primary objective of this study is to evaluate the safety of Serp-1 injection when administered in 3 daily doses to patients undergoing conventional therapy for Acute Coronary Syndrome (ACS) requiring early intervention.

DETAILED DESCRIPTION:
A total of 72 subjects will be enrolled, separated into 3 dose groups and centrally randomized in a 3:1 ratio of Serp-1 injection to placebo control.Subjects will receive Serp-1 by intravenous (IV) bolus injection daily for 3 days, at dose levels of 5.0, 15, and 50 ug/kg/dose or placebo (0.9% normal saline) added to any prescribed therapy for ACS. Serp-1 will be administered as a single IV bolus injection. The initial IV bolus dose is administered immediately preceding the PCI procedure with subsequent doses administered 24 and 48 hours later.Subjects will be evaluated for adverse events, serum inflammatory markers and restenosis rates at 6 months post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of unstable angina or NSTEMI with one or more episodes of angina in the 24 hours before hospital admission
* Scheduled for PCI

Exclusion Criteria:

* CABG within 6 months
* Acute ST elevation, eligible for thrombolysis on initial examination
* Coronary lesions with total thrombotic occlusions
* Current immunosuppressant therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse events collected until 6 months post-dose)

SECONDARY OUTCOMES:
Inflammatory marker analysis
MACE
Restenosis at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Lucas, MD, Study Director — Chief Clinical Officer- Viron Therapeutics; Jean-Claude Tardif, MD, Study Chair — Director- Montreal Heart Institute Research Centre
Locations (8):
- United States (3):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Spectrum Health, Grand Rapids, Michigan
- Canada (5):
  - Victoria Heart Institute, Vicotria, British Columbia
  - Foothills Medical Center, Calgary, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec

REFERENCES:
- [Derived] Tardif JC, L'Allier PL, Gregoire J, Ibrahim R, McFadden G, Kostuk W, Knudtson M, Labinaz M, Waksman R, Pepine CJ, Macaulay C, Guertin MC, Lucas A. A randomized controlled, phase 2 trial of the viral serpin Serp-1 in patients with acute coronary syndromes undergoing percutaneous coronary intervention. Circ Cardiovasc Interv. 2010 Dec;3(6):543-8. doi: 10.1161/CIRCINTERVENTIONS.110.953885. Epub 2010 Nov 9. PMID 21062996